CLINICAL TRIAL: NCT00235339
Title: Comparative Study of Training Modality After Myocardial Infarction; Standard Care Rehabilitation Training or Interval Treadmill Training
Brief Title: Effect of Standard Care Rehabilitation Versus Interval Treadmill Training After Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-05-01
Record Dates: First submitted 2005-10-07; First posted 2005-10-10 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Myocardial Infarction
Keywords: Oxygen Consumption; Exercise; Rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard exercise training rehabilitation at the hospital
  Interventions: Behavioral: Exercise training
- 2 (Experimental): Interval exercise training on treadmills, with high intensity
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Standard exercise training at the hospital, two times per week for twelve weeks
  Arms: 1
Behavioral: Exercise training — Interval exercise training with high intensity on treadmill. Subjects exercise two times per week for twelve weeks
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effect of the standard rehabilitation offered by three hospital rehabilitation units in Norway, one in Trondheim, one in Ålesund and one in Levanger, compared to an interval treadmill training program. The subjects participating in the study are patients with myocardial infarction. The maximal oxygen consumption of the subjects will be tested before and after the training period.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of the standard rehabilitation offered by three hospital rehabilitation units in Norway, one in Trondheim, one in Ålesund and one in Levanger, compared to an interval treadmill training program. The subjects participating in the study are patients with myocardial infarction. The maximal oxygen consumption of the subjects will be tested before and after the training period.

Primary outcome: Maximal oxygen consumption Secondary outcomes: Blood values (for endothelial function, blood lipids, etc), flow mediated dilatation, quality of life (SF 36 and MacNew), weight, BMI, heart rate fall 1 minute after stopping the maximal treadmill test.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction 2-12 weeks ago

Exclusion Criteria:

* Heart failure
* limitations to walking on a treadmill
* failure to reach a maximal pre-test(> NYHA class II)
* uncontrolled hypertension
* COPD
* pregnancy
* kidney failure (creatinin > 140)
* drug abuse
* left ventricle EF < 30%

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-10; Primary Completion 2008-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
change in maximal oxygen consumption | baseline, after intervention and at 6 months
  At baseline, following intervention and at 6 months after the intervention. An additional follow-up test will be conducted in all patients who want to participate during 2009.

SECONDARY OUTCOMES:
quality of life | baseline, after intervention and at 6 months
flow mediated dilatation | baseline, after intervention and at 6 months
  flow mediated dilatation (endothelial function)
echocardiography | baseline, after intervention and at 6 months
blood markers | baseline, after intervention and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stig A Slørdahl, Dr.med, Study Chair — National Taiwan Normal University; Trine T Moholdt, Cand.polit, Principal Investigator — National Taiwan Normal University
Locations (3):
- Norway (3):
  - Sykehuset Levanger, Levanger, Levanger
  - Ålesund Hospital, Ålesund
  - St.Olav Hospital, Trondheim

REFERENCES:
- [Result] Moholdt T, Aamot IL, Granoien I, Gjerde L, Myklebust G, Walderhaug L, Hole T, Graven T, Stolen T, Molmen-Hansen HE, Stoylen A, Skogvoll E, Slordahl SA, Wisloff U. Long-term follow-up after cardiac rehabilitation: a randomized study of usual care exercise training versus aerobic interval training after myocardial infarction. Int J Cardiol. 2011 Nov 3;152(3):388-90. doi: 10.1016/j.ijcard.2011.08.025. Epub 2011 Sep 9. No abstract available. PMID 21907424
- [Result] Moholdt T, Aamot IL, Granoien I, Gjerde L, Myklebust G, Walderhaug L, Brattbakk L, Hole T, Graven T, Stolen TO, Amundsen BH, Molmen-Hansen HE, Stoylen A, Wisloff U, Slordahl SA. Aerobic interval training increases peak oxygen uptake more than usual care exercise training in myocardial infarction patients: a randomized controlled study. Clin Rehabil. 2012 Jan;26(1):33-44. doi: 10.1177/0269215511405229. Epub 2011 Sep 21. PMID 21937520